CLINICAL TRIAL: NCT02637596
Title: Quality of Life After Intraoperative Radiofrequency Ablation of Pancreatic Cancer
Brief Title: Quality of Life After Radiofrequency Ablation of Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Jan Hlavsa, Jan Hlavsa MD, PhD, principal investigator, Brno University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT 14579-3
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RFA group (Experimental): Twenty-fourth consecutive patients with histologically proved pancreatic cancer [stage IIb (n=4), III (n=15), IV (n=5) ]underwent intraoperative RFA of primary tumor.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — After laparotomy, intraoperative IOUS quided RFA of primary tumor was performed.
  Other Names: RFA

SUMMARY:
A prospective clinical study evaluating quality of life (QoL) in pancreatic cancer patients treated with intraoperative radiofrequency ablation (RFA).

ELIGIBILITY:
Inclusion Criteria:

* histologically proved locally advanced or metastatic pancreatic cancer. Patients with histologically proved resectable pancreatic cancer with low Karnofsky index.

informed consent

Exclusion Criteria:

* cystic tumor

age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of life after RFA of pancreatic cancer | 3 years
  Quality of life will be evaluated using EORTC C 30 and pan 26 questionaire preoperatively and three months after RFA

SECONDARY OUTCOMES:
3- months perioperative morbidity and mortality | 3 years
  Three months morbidity and mortality will be evaluated using Dindo-Clavien classification

OTHER OUTCOMES:
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hlavsa, MD, PhD, Principal Investigator — Department of surgery Masaryk University Hospital Brno
Locations (1):
- Department of surgery Masaryk University Hostpital Brno, Brno, Bohunice, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Publication as manuscript